CLINICAL TRIAL: NCT02163551
Title: Respiratory Event-Related Potentials in Patients With Spinal Cord Injury: An Evaluation of Somatosensory Afferents
Brief Title: Respiratory Event-Related Potentials in Patients With Spinal Cord Injury
Status: Terminated | Type: Observational
Why Stopped: Recurrent equipment failures (used with custom EEG and ERP recording software) precluded timely data collection and analysis activities.
Sponsor: University of North Carolina, Charlotte (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Andrew Harver, Professor, University of North Carolina, Charlotte
Other Study IDs: 13-07-09
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Spinal Cord Injury
Keywords: dyspnea; respiratory sensation; event-related potentials; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Spinal Cord Injury: Participants with spinal cord injury (n = 20) will be age 30-60 years with motor complete spinal cord injuries, otherwise known as American Spinal Injury Association (ASIA) classification A or B, between the levels of C3 and T12. Patients will have to be able to breathe independently without the use of a ventilator. Subjects will be divided equally into four different injury level categories. The four categories are high tetraplegia (C3 - C5), low tetraplegia (C6-C8), high paraplegia (T1-T6), and low paraplegia (T7-T12).
- Controls: Twenty healthy age-matched adults will also participate.

SUMMARY:
Dyspnea is "a subjective experience of breathing discomfort that consists of qualitatively distinct sensations that vary in intensity". It is known that sensory information from the respiratory system activates regions of the cerebral cortex to produce the perception of dyspnea but far less is known about the neurophysiology of dyspnea than about vision, hearing, or even pain. Dyspnea likely arises from multiple nervous system sources, but the exact locations have not been well identified. Investigations of the mechanisms underlying respiratory sensations have included studies of airway anesthesia, chest wall strapping, exercise, heart-lung transplantation, hyperventilation, and opioid use. Study of the perception of breathing sensations in individuals with a spinal cord injury presents additional opportunity. The goal of the proposed project is to examine the effects of increasingly severe levels of spinal cord injury on the perception of breathing sensations in participants who are able to breathe without the use of a ventilator. The investigators hypothesize that the perception of breathing varies with the extent of somatosensory information that reaches cerebral cortex.

DETAILED DESCRIPTION:
Dyspnea is "a subjective experience of breathing discomfort that consists of qualitatively distinct sensations that vary in intensity." Dyspnea, or shortness of breath, is a common problem affecting up to half of hospitalized patients; and "shortness of breath" and "labored or difficult breathing" accounts for 3 to 4 million emergency department visits annually. Dyspnea can represent a sensation, a symptom, or an illness. Each set of experiences involves distinct sensory, perceptual, and cognitive processes, including: the detection of signals; the perception of threat or remarkable challenge; and, the construction, or mental representation, of illness. As a sensory experience dyspnea can be compared to the sensation of pain. Although labored breathing is not painful in the usual sense of the word dyspnea, like pain, is a concept varying along multiple dimensions. Like pain, dyspnea can signal the need for medical attention; but unlike pain dyspnea is a localized sensation originating in the cardiopulmonary system rather than a generalized danger signal.

Research demonstrates that sensory information from the respiratory system activates regions of the cerebral cortex to produce the perception of dyspnea but far less is known about the neurophysiology of dyspnea than about vision, hearing, or even pain. Dyspnea likely arises from multiple nervous system sources. Investigations of the mechanisms underlying respiratory sensations have included studies of airway anesthesia, chest wall strapping, exercise, heart-lung transplantation, hyperventilation, and opioid use. Study of the perception of breathing sensations in individuals with a spinal cord injury presents additional opportunity. The goal of the proposed project is to examine the effects of increasingly severe levels of spinal cord injury on the perception of breathing sensations in participants who are able to breathe without the use of a ventilator.

Afferent pathways that transmit somatosensory signals to the central nervous system (i.e., brain and spinal cord) are well described and event-related potentials have been used to measure respiratory somatosensation with high temporal resolution. Event-related potentials (ERPs) are time-locked cortical signals that are measured non-invasively from the surface of the scalp in response to brief (< 200 msec), presentations of respiratory stimuli during normal breathing. Davenport et al. first identified sensory-perceptual ERPs to inspiratory stimuli (those occurring about 50-150 msec after stimulus delivery) and Harver et al. first examined perceptual-cognitive ERPs to inspiratory stimuli (those occurring about 150-400 msec post-stimulus). Study of respiratory-related ERPs in patients with spinal cord injuries presents a rare opportunity to examine the neurophysiological mechanisms underlying the perception of breathing because the extent of somatosensory information that reaches cerebral cortex varies with level of lesion.

ELIGIBILITY:
Inclusion Criteria:

* Participants with spinal cord injury (n = 20) will be age 30-60 years with motor complete spinal cord injuries, otherwise known as American Spinal Injury Association (ASIA) classification A or B, between the levels of C3 and T12. Subjects will be divided equally into four different injury level categories. The four categories are high tetraplegia (C3 - C5), low tetraplegia (C6-C8), high paraplegia (T1-T6), and low paraplegia (T7-T12). Twenty healthy age-matched adults will also participate.

Exclusion Criteria:

* History or presence of lung disease (asthma, chronic bronchitis, etc)
* Current smoker (more than one cigarette per day the past year)
* History of traumatic brain injury, epilepsy, or seizure; using psychotropic medication of any type
* And, if patient, more than six months since spinal cord injury and clinically stable.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with spinal cord injury will participate in an initial enrollment session at Carolinas Rehabilitation. Patients will be recruited from a registry managed by Dr. Lieberman. Healthy volunteers will be recruited through e-mail solicitation for volunteers for a project examining breathing sensations distributed to faculty, students, and staff in the College of Health and Human Services.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Event-Related Potentials | Baseline, 2-3 hours
  To record event-related potentials, surface electrodes will be attached with electrode collars and paper tape. Electrodes will be positioned at Fz (frontal midline), Cz (central midline), Pz (parietal midline), 1 cm below the center of the right eye to monitor eye movements, on the right mastoid (reference site), and on the forehead (ground site).

SECONDARY OUTCOMES:
General Health Status | Baseline,1 hour
  Participants will complete general and respiratory health histories, a standardized Respiratory Disease Questionnaire, and a measure of quality of life (SF-36).

OTHER OUTCOMES:
Lung Function | Baseline, 1 hour
  Participants perform lung function testing, hold their breaths for as a long as possible, and produce maximal inspiratory and expiratory efforts against a closed airway.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Harver, PhD, Principal Investigator — University of North Carolina, Charlotte; Jesse A. Lieberman, MD, MSPH, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Spinal Cord Injury Medicine, Carolinas Rehabilitation, Charlotte, North Carolina
  - UNC Charlotte, Charlotte, North Carolina

REFERENCES:
- [Background] Parshall MB, Schwartzstein RM, Adams L, Banzett RB, Manning HL, Bourbeau J, Calverley PM, Gift AG, Harver A, Lareau SC, Mahler DA, Meek PM, O'Donnell DE; American Thoracic Society Committee on Dyspnea. An official American Thoracic Society statement: update on the mechanisms, assessment, and management of dyspnea. Am J Respir Crit Care Med. 2012 Feb 15;185(4):435-52. doi: 10.1164/rccm.201111-2042ST. PMID 22336677
- [Background] Bloch-Salisbury E, Harver A, Squires NK. Event-related potentials to inspiratory flow-resistive loads in young adults: stimulus magnitude effects. Biol Psychol. 1998 Sep;49(1-2):165-86. doi: 10.1016/s0301-0511(98)00034-9. PMID 9792492
- [Background] Harver A, Squires NK, Bloch-Salisbury E, Katkin ES. Event-related potentials to airway occlusion in young and old subjects. Psychophysiology. 1995 Mar;32(2):121-9. doi: 10.1111/j.1469-8986.1995.tb03303.x. PMID 7630976
- [Background] Bloch-Salisbury E, Harver A. Effects of detection and classification of resistive and elastic loads on endogenous event-related potentials. J Appl Physiol (1985). 1994 Sep;77(3):1246-55. doi: 10.1152/jappl.1994.77.3.1246. PMID 7836128
- [Background] Davenport PW, Friedman WA, Thompson FJ, Franzen O. Respiratory-related cortical potentials evoked by inspiratory occlusion in humans. J Appl Physiol (1985). 1986 Jun;60(6):1843-8. doi: 10.1152/jappl.1986.60.6.1843. PMID 3722053